CLINICAL TRIAL: NCT02485067
Title: Multicenter, Randomized, Double-blind, Parallel, Active Control, Phase III Clinical Study to Assess the Efficacy and Safety of THVD-201 in Patients With Overactive Bladder Including an Open-label, Extension Study
Brief Title: Clinical Study to Assess the Efficacy and Safety of THVD-201 in Patients With OAB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THVD-201_OAB_III_2014
Record Dates: First submitted 2015-06-12; First posted 2015-06-30 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Tolterodine (Detrusitol); Pilocarpine
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- THVD-201 (Experimental): 1. Treatment period(12 weeks)
  1. Double dummy(A+B) A. THVD-201: capsule B. Placebo(For Detrusitol 2mg tablet)
  2. One capsule and One tablet bid on an empty stomach
  2. Open-label extension period(An additional 12 weeks)
  1. Regardless of the previous type of arm, all patients only take THVD-201 during this period.
  2. One capsule bid on an empty stomach
  Interventions: Drug: THVD-201; Drug: Placebo(For Detrusitol 2mg tablet)
- Tolterodine (Detrusitol) (Active Comparator): 1. Treatment period(12 weeks)
  1. Double dummy(A+B) A. Placebo(For THVD-201): capsule B. Detrusitol 2mg tablet
  2. One capsule and One tablet bid on an empty stomach
  2. Open-label extension period(An additional 12 weeks)
  1. Regardless of the previous type of arm , all patients only take THVD-201 during this period.
  2. One capsule bid on an empty stomach
  Interventions: Drug: THVD-201; Drug: Placebo(For THVD-201); Drug: Detrusitol 2mg tablet

INTERVENTIONS:
Drug: THVD-201 — Combination of Tolterodine 2mg and Pilocarpine 9mg
Drug: Placebo(For THVD-201)
  Arms: Tolterodine (Detrusitol)
Drug: Detrusitol 2mg tablet — Tolterodine 2mg
  Arms: Tolterodine (Detrusitol)
Drug: Placebo(For Detrusitol 2mg tablet)
  Arms: THVD-201

SUMMARY:
The primary purpose of this study is to assess the efficacy and safety of THVD-201(Combination of tolterodine and pilocarpine) in patients with Overactive bladder during the period of treatment, 12 weeks.

This study also includes an open label extension period of an additional 12 weeks following the treatment to assess long-term efficacy and safety of THVD-201 in patients with Overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* 20 - 85 years
* History of OAB (pure urge or mixed urinary incontinence with predominant urge incontinence) for ≥ 6 months.
* In the case of females, at least 2 years has passed since menopause. Or all pre-menopausal female subjects must have been using a highly effective method of birth control during the study. Subject of childbearing potential must have had a negative pregnancy test prior to enrollment.

Exclusion Criteria:

* Predominate stress incontinence, insensate incontinence (those incapable of distinguishing discrete incontinence episodes) and overflow incontinence, as major reason for urine loss or urinary frequency as determined by the investigator.
* History of neurogenic bladder.
* PVR > 200mL
* History of clinically significant renal disease or estimated creatinine clearance defined by Cockcroft and Gault formula < 30 mL/min.
* History of malignant tumor within the past 5 years.
* History or presence of tachyarrhythmia or cardiac disease that in the opinion of the investigator might have confounded the results of the study or posed additional risk to the subject. Subjects who had a value for QTc > 450 msec at the Screening visit.
* Patient with asthma
* PSA ≥ 10 ng/mL in male who is 50 years and over.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Mean daily micturition frequency | 12 weeks
  The change of Mean daily micturition frequency between 0 and 12 weeks
ADR Incidence of Dry mouth | 12 weeks

SECONDARY OUTCOMES:
Mean daily micturition frequency | 24 weeks
  The change of Mean daily micturition frequency between 0 and 24 weeks
Mean daily Incontinence frequency(12 weeks) | 12 weeks
  The change of Mean daily Incontinence frequency between 0 and 12 weeks
Mean daily Incontinence frequency(24 weeks) | 24 weeks
  The change of Mean daily Incontinence frequency between 0 and 24 weeks
Mean daily Urgency frequency(12 weeks) | 12 weeks
  The change of Mean daily Urgency frequency between 0 and 12 weeks
Mean daily Urgency frequency(24 weeks) | 24 weeks
  The change of Mean daily Urgency frequency between 0 and 24 weeks
Mean daily Nocturia frequency(12 weeks) | 12 weeks
  The change of Mean daily Nocturia frequency between 0 and 12 weeks
Mean daily Nocturia frequency(24 weeks) | 24 weeks
  The change of Mean daily Nocturia frequency between 0 and 24 weeks
Mean daily Micturition volume(12 weeks) | 12 weeks
  The change of Mean daily Micturition volume between 0 and 12 weeks
Mean daily Micturition volume(24 weeks) | 24 weeks
  The change of Mean daily Micturition volume between 0 and 24 weeks
Score of OAB-SS questionnaire(12 weeks) | 12 weeks
  The change of the Score between 0 and 12 weeks
Score of OAB-SS questionnaire(24 weeks) | 24 weeks
  The change of the Score between 0 and 24 weeks
Score of OAB-q questionnaire(12 weeks) | 12 weeks
  The change of the Score between 0 and 12 weeks
Score of OAB-q questionnaire(24 weeks) | 24 weeks
  The change of the Score between 0 and 24 weeks
VAS score of dry mouth symptom(12 weeks) | 12 weeks
  The change of the Score between 0 and 12 weeks
VAS score of dry mouth symptom(24 weeks) | 24 weeks
  The change of the Score between 0 and 24 weeks
Score of Xerostomia Inventory questionnaire(12 weeks) | 12 weeks
  The change of the Score between 0 and 12 weeks
Score of Xerostomia Inventory questionnaire(24 weeks) | 24 weeks
  The change of the Score between 0 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Sung Lee, Principal Investigator — Samsung Medical Center (SMC)
Locations (16):
- South Korea (16):
  - Inje University Busan Paik Hospital, Busan
  - Dankook University Hospital, Cheonan
  - Chonnam National University Hospital, Gwangju
  - Pusan National University Hospital, Pusan
  - Bundang Cha Medical center, Seongnam
  - Ajou University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Cheil General Hospital, Seoul
  - Gachon University Gil Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Bucheon ST. Mary's Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul